CLINICAL TRIAL: NCT07291115
Title: Analysis of the Physical Fitness Development Trajectory of Children and Adolescents With Severe Intellectual Disabilities in Orphanages: A Three-Year Longitudinal Follow-Up Study
Acronym: SID-FIT
Status: Completed | Type: Observational
Sponsor: Xili Wen (Other)
Responsible Party: Sponsor-Investigator, Xili Wen, Ph.D Student, Shanghai University of Sport
Organization: Shanghai University of Sport (Other)
Other Study IDs: Fitness Development Trajectory
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Severe Intellectual Disability; Intellectual Disability
Keywords: Severe intellectual disability; Physical fitness; Longitudinal study; Body mass index; Motor fitness
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orphanage Cohort: This cohort includes all children and adolescents with severe intellectual disabilities who were permanent residents of the participating state-run orphanages in Kaifeng, Zhengzhou, Wuhan, and Hohhot, China. Participants were 7-18 years old at baseline and were followed prospectively for three years with repeated physical fitness assessments. No experimental intervention was introduced; all participants continued to receive usual institutional care and routine school-based physical education.
  Interventions: Other: Usual institutional care and school-based physical education

INTERVENTIONS:
Other: Usual institutional care and school-based physical education — Participants receive the usual institutional care and routine school-based physical education provided by their orphanages. The study does not introduce any experimental intervention; physical fitness is measured repeatedly over three years under real-world conditions.

SUMMARY:
This observational cohort study was designed to describe how physical fitness changes over time in children and adolescents with severe intellectual disabilities living in orphanages in China. A total of 132 participants aged 7-18 years were recruited from four state-run orphanages and followed prospectively for three years. At baseline and every 3 months thereafter (12 assessments in total), trained assessors measured body mass index and simple field-based fitness tests, including beanbag throwing for upper limb strength, sit-ups for core strength, standing long jump for lower limb explosive strength, and one-leg standing for static balance.

The main aim of the study is to characterize the long-term trajectories of physical fitness in this highly vulnerable population and to examine whether patterns of change differ by age group (children 7-12 years vs adolescents 13-18 years) and by sex. The findings are intended to provide evidence to guide physical education programming and health management strategies for children and adolescents with severe intellectual disabilities living in institutional care settings.

DETAILED DESCRIPTION:
Background and Rationale Children and adolescents with severe intellectual disabilities (SID) often present with marked limitations in motor skills, low levels of physical activity, and elevated risk of secondary health problems. Those living in orphanages represent an especially vulnerable group, as they frequently have limited access to individualized physical education and health promotion programs. However, there is little longitudinal evidence describing how physical fitness develops over time in this population, and whether trajectories differ by age or sex. Understanding these patterns is essential for designing tailored interventions and for allocating rehabilitation and educational resources within institutional care settings.

Study Design and Objectives This study is a prospective, multi-site, observational cohort. The overarching objective is to analyze three-year development trajectories of physical fitness among children and adolescents with SID residing in orphanages. Specific objectives are: (1) to describe longitudinal changes in body mass index (BMI), upper limb strength, core strength, lower limb explosive strength, and static balance over 12 measurement occasions; and (2) to compare these trajectories between age groups (children 7-12 years vs adolescents 13-18 years) and between boys and girls. No experimental intervention is introduced; all participants continue to receive usual institutional care and routine school-based physical education.

Setting and Participants Participants were recruited from four state-run orphanages located in Kaifeng and Zhengzhou (Henan Province), Wuhan (Hubei Province), and Hohhot (Inner Mongolia), China. At baseline, eligible participants were 7-18 years old, had a clinical diagnosis of severe intellectual disability according to national standards, and were permanent residents of the participating orphanages. Children and adolescents with acute or unstable medical conditions that would preclude participation in basic fitness testing, or with other contraindications judged by institutional physicians, were excluded. Written informed consent was obtained from legal guardians or institutional representatives in accordance with local regulations and the ethics approval.

Assessments and Outcome Measures

Data collection started in March 2021 (T1) and continued for three years with follow-up assessments every 3 months (approximately June, September, and December each year) until March 2024, yielding 12 planned measurement time points. At each assessment, trained physical education teachers or research staff conducted standardized measurements:

Body mass index (BMI, kg/m²), calculated from height and weight.

Upper limb strength, assessed by beanbag throwing distance (meters).

Core strength, assessed by the number of correctly performed sit-ups within 1 minute.

Lower limb explosive strength, assessed by standing long jump distance (meters).

Static balance, assessed by one-leg standing time (seconds).

These measures constitute the primary and secondary outcome variables for the study. Sociodemographic characteristics (age, sex) and basic clinical information were also recorded at baseline.

Planned Data Analysis The primary analytic approach is to use generalized estimating equations (GEE) to model longitudinal changes in each fitness indicator across the 12 repeated assessments, accounting for within-subject correlation and unbalanced follow-up. Time (measurement occasion), age group at baseline (children vs adolescents), sex, and their interactions are included as predictors to estimate developmental trajectories and group differences. Analyses are conducted on the full cohort of 132 participants who contributed at least one measurement, consistent with an intention-to-follow principle for observational data.

Ethical Considerations and Status The protocol was reviewed and approved by the Ethics Committee of the Shanghai University of Physical Education and Sport (Approval No. 102772020RT054). All assessments were conducted during regular school hours using low-risk, field-based tests appropriate for children and adolescents with SID. Data collection has been completed, and this record provides a transparent description of the study procedures and analysis plan.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of severe intellectual disability according to national or institutional diagnostic standards.

Aged 7 to 18 years at baseline.

Permanent resident of one of the participating state-run orphanages in Kaifeng, Zhengzhou, Wuhan, or Hohhot, China.

Able, with assistance if needed, to follow simple instructions and to attempt the basic physical fitness tests used in the study (height and weight, beanbag throwing, sit-ups, standing long jump, and one-leg standing).

Written informed consent provided by the legal guardian or institutional representative in accordance with local regulations and the ethics approval.

Exclusion Criteria:

Presence of an acute or unstable medical condition (e.g., severe cardiopulmonary disease, uncontrolled epilepsy, acute musculoskeletal injury) that would preclude safe participation in basic physical fitness testing.

Any other condition or behavioural problem that, in the judgement of the institutional physician or investigators, would make participation unsafe or seriously interfere with completion of the assessments.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 7-18 years with severe intellectual disabilities who are permanent residents of four state-run orphanages located in Kaifeng and Zhengzhou (Henan Province), Wuhan (Hubei Province), and Hohhot (Inner Mongolia), China. All eligible residents meeting the inclusion criteria were invited to participate and were followed prospectively for three years with repeated physical fitness assessments. No healthy controls were included.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in body mass index (BMI) | From baseline (March 2021) to 36 months (March 2024), assessed at 12 time points (every 3 months).
  Body mass index (BMI, kg/m²) measured at each assessment using standardized height and weight measurements. BMI values will be analyzed using generalized estimating equations (GEE) to estimate the three-year trajectory and to compare patterns of change by age group (children 7-12 years vs adolescents 13-18 years) and by sex.
Longitudinal change in upper limb strength (beanbag throwing distance) | From baseline (March 2021) to 36 months (March 2024), assessed at 12 time points (every 3 months).
  Upper limb strength assessed by beanbag throwing distance (meters) at each assessment. The best of two trials will be recorded. Generalized estimating equations (GEE) will be used to model three-year trajectories and to compare patterns of change by age group and sex.
Longitudinal change in core strength (sit-ups) | From baseline (March 2021) to 36 months (March 2024), assessed at 12 time points (every 3 months).
  Core strength assessed by the number of correctly performed sit-ups in 1 minute at each assessment. Generalized estimating equations (GEE) will be used to model three-year trajectories and to compare patterns of change by age group and sex.
Longitudinal change in lower limb explosive strength (standing long jump distance) | From baseline (March 2021) to 36 months (March 2024), assessed at 12 time points (every 3 months).
  Lower limb explosive strength assessed by standing long jump distance (meters) at each assessment. The best of two trials will be recorded. Generalized estimating equations (GEE) will be used to model three-year trajectories and to compare patterns of change by age group and sex.
Longitudinal change in static balance (one-leg standing time) | From baseline (March 2021) to 36 months (March 2024), assessed at 12 time points (every 3 months).
  Static balance assessed by one-leg standing time (seconds) at each assessment. The best performance will be recorded. Generalized estimating equations (GEE) will be used to model three-year trajectories and to compare patterns of change by age group and sex.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Sport, School of Physical Education and Training, Shanghai, Ph.d, China

IPD SHARING:
Plan to Share IPD: No